CLINICAL TRIAL: NCT05705609
Title: The Effect of Mandala Art Therapy on Blood Glucose Level, Mood and Anxiety in Pregnant Women With Abnormal OGTT: A Randomized Controlled Study
Brief Title: The Effect of Mandala Art Therapy on Pregnant Women With Abnormal OGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: İnönü University (Unknown)
Responsible Party: Principal Investigator, ESRA GUNEY, PhD, PhD, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3679
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related
Keywords: Pregnant Women; Oral Glucose Tolerance Test; Anxiety; Affect
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial conducted with experimental and control groups.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala art therapy (Experimental): Mandala art therapy applied group
  Interventions: Other: Mandala art therapy
- Standard of care (No Intervention): group without Mandala art therapy

INTERVENTIONS:
Other: Mandala art therapy — A mandala is a geometric configuration of symbols. In various spiritual traditions, mandalas may be employed for focusing attention of practitioners and adepts, as a spiritual guidance tool, for establishing a sacred space and as an aid to meditation and trance induction. Mandalas are used effectively in the field of art therapy. The possibility of using mandala in all age groups has contributed to the treatment process of different diseases and disorders, and its effectiveness has been presented to the scientific world with many researches around the globe. As a result of using mandala as an art therapy in adults, mandala has been used both in the treatment of psychiatric disorders and has been a tool used to observe the effects of the treatments. Art therapy which included drawing mandala, significantly reduced the severity of trauma symptoms in individuals with anxiety disorders and post-traumatic stress disorder.
  Arms: Mandala art therapy

SUMMARY:
The goal of this interventional study is to learn about determine the effect of mandala art therapy on blood glucose level, mood and anxiety in pregnant women with abnormal oral glucose tolerance test (OGTT) value. The main questions it aims to answer are:

* Does mandala art therapy affect the mood of pregnant women?
* Does mandala art therapy affect the anxiety level of pregnant women?

After measuring fasting plasma glucose and drinking oral glucose by the hospital staff in the experimental group in the outpatient clinic, after the 1st and 2nd hour measurements, a total of 2 individual mandala activities (Mandala training certificate was obtained by Dr. Lecturer Esra KARATAŞ OKYAY) will be performed by the researcher.

DETAILED DESCRIPTION:
The goal of this interventional study is to learn about determine the effect of mandala art therapy on blood glucose level, mood and anxiety in pregnant women with abnormal oral glucose tolerance test (OGTT) value.

Pregnant women who apply to Malatya Training and Research Hospital gynecology outpatient clinics to have OGTT and meet the criteria will be invited to the study. The women will be informed about the method to be followed in the research, the voluntary information form will be read to those who want to participate in the research, and their verbal and written permissions will be obtained. Before Mandala art therapy, a personal information form, State Meta-Mood Scale (SMMS) and State Trait Anxiety Scale (STAI) will be applied to pregnant women in both groups. All blood collection and OGTT procedures for pregnant women in the experimental and control groups will be performed by hospital staff in line with hospital procedures. After measuring fasting plasma glucose and drinking oral glucose by the hospital staff in the experimental group in the outpatient clinic, after the 1st and 2nd hour measurements, a total of 2 individual mandala activities (Mandala training certificate was obtained by one of researcher Esra KARATAŞ OKYAY) will be performed by the researcher. The blood glucose levels of the pregnant woman at the time of measurement will be recorded from the patient records. As a post-test, the State Meta-Mood Scale (SMMS) and state anxiety scale will be applied again. Any procedure other than routine care will not be applied to the pregnant women in the control group. Likewise, the blood glucose levels of the pregnant woman at the time of measurement will be recorded from the patient records. As a post-test, the State Meta-Mood Scale (SMMS) and StateTrait Anxiety Scale (STAI) will be applied again.

ELIGIBILITY:
Inclusion Criteria:

* at 24-28 weeks of gestation,
* OGTT will be done,
* Those who have not received mandala art therapy training before,
* Does not have a physical problem that will prevent creating a mandala,
* Actively using their hands
* No communication problem
* Pregnant women without learning problems were included in the sample

Exclusion Criteria:

* Any problems diagnosed in pregnancy (such as oligohydramnios, preeclampsia, heart disease, diabetes, placenta previa)
* Pregnant women diagnosed with gestational diabetes
* Pregnant women in their first term were not included in the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Anxiety scores | at 1st hours after OGTT
  StateTrait Anxiety Scale (STAI): The highest score from the scale is 80, the lowest score is 20. Higher STAI-I scores indicate higher state anxiety levels
Anxiety scores | at 2nd hours after OGTT
  StateTrait Anxiety Scale (STAI): The highest score from the scale is 80, the lowest score is 20. Higher STAI-I scores indicate higher state anxiety levels

SECONDARY OUTCOMES:
Mood scores | at 1st hours after OGTT
  State Meta-Mood Scale: The highest score from the scale is 32, the lowest score is 8. High scores indicate high mood
Mood scores | at 2nd hours after OGTT
  State Meta-Mood Scale: The highest score from the scale is 32, the lowest score is 8. High scores indicate high mood

CONTACTS AND LOCATIONS:
Overall Officials: ESRA GÜNEY, PhD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared.

REFERENCES:
- [Result] Kim H, Kim S, Choe K, Kim JS. Effects of Mandala Art Therapy on Subjective Well-being, Resilience, and Hope in Psychiatric Inpatients. Arch Psychiatr Nurs. 2018 Apr;32(2):167-173. doi: 10.1016/j.apnu.2017.08.008. Epub 2017 Aug 24. PMID 29579508
- See also: Reference link — https://pubmed.ncbi.nlm.nih.gov/29579508/
- Available data/document: Informed Consent Form: Kim H, Kim S, Choe K, Kim JS — https://pubmed.ncbi.nlm.nih.gov/29579508/ — web site is provided